CLINICAL TRIAL: NCT01652859
Title: An Open-label, Randomized, Balanced, Crossover Bioequivalence Study to Compare Two 2 mg/ml Liposomal Amphotericin B Injections in Healthy Subjects
Brief Title: An Bioequivalence Study to Compare Two 2 mg/ml Liposomal Amphotericin B Injections in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Taiwan Liposome Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: TLC166.2
Record Dates: First submitted 2012-07-20; First posted 2012-07-30 (Estimated); Last update posted 2013-11-27 (Estimated); Status verified 2013-11

CONDITIONS: Normal Healthy Subjects
MeSH Terms: interventions — liposomal amphotericin B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Liposomal Amphotericin B (Experimental): Generic drug
  Interventions: Drug: Liposomal Amphotericin B
- AmBisome (Active Comparator): RLD
  Interventions: Drug: AmBisome

INTERVENTIONS:
Drug: Liposomal Amphotericin B
  Arms: Liposomal Amphotericin B
Drug: AmBisome
  Arms: AmBisome

SUMMARY:
The 2 × 2 crossover designed study is to evaluate the bioequivalence of two different liposomal amphotericin B injections after single IV infusion at the same dose in normal healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be adults (> 20 years old) in good health on the basis of medical history, physical examination, electrocardiogram, chest X-ray, and routine laboratory evaluations.
2. Vital signs (after 3 minutes resting in a upright position) which are within the following ranges: Ear body temperature between 35.0-37.5 °C. Systolic blood pressure, 90-140 mm Hg. Diastolic blood pressure, 50-90 mm Hg. Pulse rate, 50-90 bpm
3. Fasting blood glucose < 100 mg/dL.
4. Body weight must be above 50 kg for men and 45 kg for women and within 20% of ideal body weight.
5. Negative urine drug screen at clinic check-in before each dosing
6. Able to sign informed consent prior to study.
7. Able to communicate well with the investigator and comply with the requirements of the study.
8. Pregnancy tests (female only): negative reaction

Exclusion Criteria:

1. Use of any prescription or over the counter medication within 14 days prior to investigational products administration; with the exception of acetaminophen (not more than 2 g/day) or vitamins.
2. A plan to take concomitant medications while enrolled in the study, with the exception of acetaminophen (not more than 2 g/day) or vitamins.
3. Presence of any acute or chronic medical condition within 2 weeks prior to investigational products administration, including but not limited to: hepatic, gastrointestinal, renal, hematologic (including coagulation), pulmonary, neurologic, respiratory, endocrine, or cardiovascular system abnormalities; psychiatrical disease including major psychiatric disorders (e.g., schizophrenia, bipolar disorder); acute infection; or other conditions that would interfere with the absorption, distribution, metabolism, or excretion of drugs. Evidence of impaired renal function as indicated by clinically significant abnormal creatinine or BUN values or abnormal urinary constituents (e.g., albuminuria) as judged by the investigator. Evidence of liver disease, hepatitis B, hepatitis C or liver injury as indicated by an clinically significant abnormal liver function profile such as GOT, GPT, g-GT, alkaline phosphatase, serum bilirubin, HBs Ag, or HCV Ab as judged by the investigator.
4. Hemoglobin less than 12 g/dL
5. Participation in any clinical investigation within 2 months or 5 half-lives, whichever is longer, prior to investigational products administration.
6. Donation or loss of more than 500 mL blood within 3 months prior to investigational products administration.
7. Subject is known for HIV infected.
8. Known allergy or hypersensitivity to amphotericin B or its analogs.
9. History of drug or alcohol abuse within 12 months prior to investigational products administration ; current consumption of alcohol in excess of 28 units/week (one unit is 6 oz of beer, ½ oz of hard liquor, or 2 oz of wine)
10. Subjects who, in the opinion of the investigator, should not participate in the study or may not be capable of following the study schedule for any reason.
11. Consumption of more than 36 to 40 oz (1.1-1.2 L) of caffeine-containing beverages per day
12. Consumption of any products containing grapefruit in the 3 days before clinic check-in.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2012-02; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
The bioequivalence of two different liposomal amphotericin B injections | 14 days
  90% CI of Cmax and AUCinf of Liposomal and non-liposomal Amphotericin B between Ambil and AmBisome within 80.00%~125.00%.

REFERENCES:
- [Derived] Adler-Moore JP, Gangneux JP, Pappas PG. Comparison between liposomal formulations of amphotericin B. Med Mycol. 2016 Mar;54(3):223-31. doi: 10.1093/mmy/myv111. Epub 2016 Jan 14. PMID 26768369